CLINICAL TRIAL: NCT05367752
Title: Short-term Effects of Myofascial Release With TENS Conductive Glove in Pain, Range of Motion and Functional Disability in Adults With Neck Myofascial Syndrome: A Randomized Clinical Trial Study
Brief Title: Effects of MR With TENS Conductive Glove in Adults With Neck Myofascial Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Hellenic University (Other)
Responsible Party: Principal Investigator, Dimitrios Lytras, Dimitrios Lytras PT, PhD, Senior Lecturer of Physiotherapy, International Hellenic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-03/2022
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Neck Pain
Keywords: Neck Pain; Myofascial trigger points; Myofascial release; Transcutaneous electrical nerve stimulation; Physiotherapy
MeSH Terms: conditions — Neck Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: An assessor-blind randomized control trial with a duration of three weeks and a one-month follow up will be performed in 80 adults with neck pain due to the presence of trigger points on the upper part of trapezius muscle. The participants will be allocated into four groups of 20 persons each (three intervention groups and one control group). In the first group, a combination therapy of myofascial release with conductive TENS gloves will be applied, in the second group the same protocol of myofascial release without conductive gloves, in the third group a high frequency (conventional) TENS, and the fourth group will get placebo TENS with the device closed. All participants will follow a total of six treatments over a period of three weeks.
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor) Assessor-blind randomized control trial. A masked assessor conducted the measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: Myofascial release with TENS conductive glove (Experimental): Participants allocated to this group received six sessions of a myofascial release protocol with a TENS conductive glove applying a TENS current of 120Hz frequency through an electrotherapy device.
  Interventions: Other: Myofascial release with TENS conductive glove
- Group 2: Myofascial release without TENS conductive glove (Experimental): Participants allocated to this group received the same myofascial release protocol with group 1 without the TENS conductive glove.
  Interventions: Other: Myofascial release without TENS conductive glove
- Group 3: Conventional TENS (Experimental): Participants allocated to this group received the application of a conventional TENS current.
  Interventions: Other: Conventional TENS
- Control: Sham TENS (Active Comparator): Participants allocated to this group received the same TENS treatment with group 3, but with the current intensity set to zero to ensure that they received no current.
  Interventions: Other: Sham TENS

INTERVENTIONS:
Other: Myofascial release with TENS conductive glove — Before each MR session, light massage and stretching was applied for five minutes as preparation for the manipulations. The massage included the effleurage technique followed by petrissage and kneading on the cervical and thoracic areas (on the upper three parts of the trapezius muscle, in the suboccipital area, and on the paraspinal cervical muscles). Stretching was applied to the following muscles: upper part of the trapezius, levator scapulae, and the sternocleidomastoid muscle.
  Upper trapezius myofascial release, unilateral gross stretch, vertical gross stretch, focused stretch, cranial base myofascial release, gross release of the sternocleidomastoid muscle, and release of the suprahyoid and infrahyoid muscles.
  Arms: Group 1: Myofascial release with TENS conductive glove
Other: Myofascial release without TENS conductive glove — Before each MR session, light massage and stretching was applied for five minutes as preparation for the manipulations. The massage included the effleurage technique followed by petrissage and kneading on the cervical and thoracic areas (on the upper three parts of the trapezius muscle, in the suboccipital area, and on the paraspinal cervical muscles). Stretching was applied to the following muscles: upper part of the trapezius, levator scapulae, and the sternocleidomastoid muscle.
  Upper trapezius myofascial release, unilateral gross stretch, vertical gross stretch, focused stretch, cranial base myofascial release, gross release of the sternocleidomastoid muscle, and release of the suprahyoid and infrahyoid muscles.
  Arms: Group 2: Myofascial release without TENS conductive glove
Other: Conventional TENS — Two 40*50mm silicone electrodes were placed with the negative electrode on the trigger point of the trapezius muscle and the positive one on the acromion. The current frequency was 120Hz and pulse duration 80ms for 30 minutes. This protocol has been proposed by Ebadi et al. (2021)
  Arms: Group 3: Conventional TENS
Other: Sham TENS — Two 40*50mm silicone electrodes were placed with the negative electrode on the trigger point of the trapezius muscle and the positive one on the acromion. The current frequency was 120Hz and pulse duration 80ms for 30 minutes. This protocol has been proposed by Ebadi et al. (2021)
  Arms: Control: Sham TENS

SUMMARY:
Myofascial neck syndrome has a high incidence in the general population and is characterized by the presence of painful trigger points in the neck muscles. Both the application of manual techniques such as myofascial release and the application of TENS currents to the painful points of the neck muscles have been proven to help reduce pain and improve the range of motion of the neck. 80 adults who will present at least one trigger point in the upper trapezius muscle will be randomly divided into four groups. In the first group, a combination therapy of myofascial release with conductive TENS glove will be applied, in the second group the same protocol of myofascial release without conductive glove, in the third group a high frequency (conventional) TENS, and the fourth group will get placebo TENS with the device closed. All participants will follow a total of six treatments over a period of three weeks with a follow-up after one month. The following will be evaluated before and after the intervention, as well as in the one-month follow-up: pain with the visual analog scale (VAS pain), Pressure Pain Threshold (PPT) in the upper trapezius muscle with a digital algometer, range of motion (ROM) of the neck with a goniometer, and functional ability with the "Neck Disability Index" (NDI) questionnaire.

DETAILED DESCRIPTION:
Background: Myofascial neck syndrome has a high incidence in the general population and is characterized by the presence of painful trigger points in the neck muscles. Both the application of manual techniques such as myofascial release (MR) and the application of transcutaneous electrical nerve stimulation (TENS) currents to the painful points of the neck muscles have been proven to help reduce pain and improve the range of motion of the neck.

Aim: To study the efficacy of the combination of MR and the simultaneous application of TENS currents in the painful points of the upper part of the trapezius muscle. The myofascial release protocol will be applied with a conductive glove, which will be connected to a TENS device so that the physiotherapist's hand can be used simultaneously as a mobile electrode.

Method: 80 adults who will present at least one trigger point in the upper trapezius muscle will be randomly divided into four groups. In the first group, a combination therapy of MR with a TENS conductive glove will be applied, in the second group the same protocol of myofascial release without conductive glove, in the third group a high frequency (conventional) TENS, and the fourth group will get placebo TENS with the device closed. All participants will follow a total of six treatments over a period of three weeks with a follow-up after one month. The following will be evaluated before and after the intervention, as well as in the one-month follow-up: pain with the visual analog scale (VAS pain), Pressure Pain Threshold (PPT) in the upper trapezius muscle with a digital algometer, range of motion (ROM) of the neck with a goniometer, and functional disability with the "Neck Disability Index" (NDI) questionnaire. For the statistical analysis of the results, a two-way ANOVA with repeated measurements will be applied.

Expected results: The combination protocol proposed in this clinical study combines the beneficial effects of TENS with the benefits of MR. For this reason, this combination is expected to be more effective than their individual application in improving the clinical picture of adults with myofascial neck syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one trigger point in the upper part of the trapezius muscle
* Age range 22-60 years
* Scoring 10% or higher on the Neck Disability Index
* Scoring of 20mm or more on the Visual Analogue Scale of pain at initial evaluation
* Written consent to participate in the study

Exclusion Criteria:

* History of acute neck injury
* Sensory disorders in the neck area
* Diagnosis with a serious illness (cancer, severe osteoporosis, infectious or inflammatory processes, fractures, congenital anomalies)

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Changes in neck pain intensity with visual analogue scale (VAS) | pre-treatment, week: 1, 3, 7
  VAS is a card with an uncalibrated scale ranging from 0-100 mm on the one side (with zero representing no pain and 100 representing the worst pain in life) with each millimeter representing one pain level. The patient subjectively estimated his or her pain level by marking a vertical line on the uncalibrated scale between zero and one hundred. Then the exact value of pain intensity could be obtained with a single ruler. Hence, the higher the value, the more intense the pain. VAS is widely used as it is easy to implement and is characterized by good psychometric properties.
Changes in Pressure Pain threshold with pressure algometry | pre-treatment, week: 1, 3, 7
  Pressure pain threshold (PPT) is defined as the minimal amount of pressure that produces pain. PPT was assessed by a digital algometer. Pressure pain threshold was assessed over the upper border of the trapezius muscle halfway between the midline and the lateral border of the acromion. The metal rod of the algometer was placed vertically on the site and the examiner applied gradually increasing pressure at a rate of 1Kg/s. PPT was calculated in kg/cm2.
Changes in functional capacity with the Greek Version of Neck disability index questionnaire | pre-treatment, week: 1, 3, 7
  Changes in functional capacity with the Greek Version of Neck disability index questionnaire It is a self-reported ten-item scale. Each item assesses different neck pain complaints. Most of the items are related to restrictions in activities of daily living, and each item is expressed by 6 different assertions in the range 0-5, with 0 indicating no disability and 5 indicating the highest disability. The total score ranges from 0 to 50. Disability Index (NDI) has sufficient support in the literature, being the most commonly used to report neck pain.
Changes in Cervical Range of Motion with bubble inclinometers and a universal goniometer | pre-treatment, week: 1, 3, 7
  Cervical active range of motion was measured with 2 bubble inclinometers. One was placed on the top of the head and the second on the spinous process of C7.Active cervical flexion, extension and side bending range of motion were assessed with participants sitting in upright position. Range of motion was measured in degrees. To measure the right and left range of flexion, a long universal goniometer will be placed at the top of the head. The arms of the goniometer will be positioned in such a way that they form a right angle with each other. One arm should face forward, while the second should look to the side towards the side of the turn to be made by the examinee, so that the goniometer reading at the beginning of the measurement is 90°. The patient will then make a turn while the examiner follows the movement without displacing the center of the goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Paris Iakovidis, PhD, Study Director — International Hellenic University
Locations (1):
- Department of Physiotherapy, Faculty of Health Sciences International Hellenic University, Thessaloniki, Sindos Thessaloníki, Greece

IPD SHARING:
Plan to Share IPD: No